CLINICAL TRIAL: NCT02783092
Title: A Double-blind, Randomized Placebo-controlled Trial to Evaluate Efficacy and Safety of Cannabidiol as an add-on Therapy for Treatment in Refractory Epileptic Crisis in Children and Adolescents
Brief Title: A Double-Blind Trial to Evaluate Efficacy and Safety of Cannabidiol as an add-on Therapy for Treatment in Refractory Epilepsy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antonio Waldo Zuardi (Other)
Collaborators: Prati Donaduzzi & Cia Ltda (Industry)
Responsible Party: Sponsor-Investigator, Antonio Waldo Zuardi, MD, PhD, Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBD-PRATI-USP_01
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Concentration unit: 200mg/ml; 5 - 25 mg/Kg/day ; Oral solution
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Oral solution of cannabidiol 200 mg / mL dissolved in corn oil. Titration period: 5 mg / kg / day up to 25 mg / kg / day. Maintenance period: highest dose obtained during the titration period (maximum of 25 mg/kg / day)
  Other Names: CBD
  Arms: Cannabidiol
Drug: Placebo — The placebo will be an oral solution of corn oil. Titration period: 5 mg / kg / day up to 25 mg / kg / day. Maintenance period: highest dose obtained during the titration period (maximum of 25 mg/kg / day)
  Other Names: PLC
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of the adjuvant use of cannabidiol administered twice daily in doses of 5-25 mg/kg/day through the proportion of responsive patients; that is, participants with at least 50% decrease in the frequency of epileptic seizures in the last month of the trial relative to baseline (pretreatment with AEDs only).

Primary end point(s): Rate of responsive patients; that is, participants with at least 50% decrease in the frequency of epileptic seizures in the last month of the trial relative to baseline (pretreatment with AEDs only).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 2 years to 18 years.
* Diagnosis of treatment-resistant epilepsy according to the criteria of the International League Against Epilepsy (ILAE) (Kwan et al., 2010).
* Participants with at least 4 epileptic seizures with intervals no longer than 21 days.
* In treatment with up to 3 AEDs concomitantly and at stable doses for at least 1 month before the baseline assessment and expected to remain stable during the period of the trial. Vagus nerve stimulation (VNS) will be considered as an AED.
* Availability of a legal guardian able to follow the protocol (e.g., understand and fill up diaries) and visitation and medication schemes, according to the decision of the investigator.
* Availability of brain neuroimaging exams (magnetic resonance or computed tomography) collected within the last 5 years.
* No significant comorbid conditions, according to medical decision, to other criteria in this Protocol, and to additional assessments: medical records, blood pressure, heart rate, and temperature measures, physical exam, ECG, EEG, and laboratory tests.
* Women in reproductive age may be included as long as they are sexually abstinent or using effective contraceptive methods.
* Participants and their legal guardians, when applicable, must sign an informed consent form approved by the local ethics committee.

Exclusion Criteria:

* Occurrence of simple partial seizures (preserved consciousness) only, with no motor symptomatology.
* History or presence of pseudoseizures.
* History of suicide attempt.
* History of major depression.
* Pregnancy.
* Drug use.
* Hypertension.
* Participants with severe dysphagia and no gastric or nasogastric tubes.
* Current treatment with drugs that may significantly affect the metabolism of CBD, except AEDs if stable for at least 1 month before the screening interview.
* Presence of any clinical or neuroimaging finding suggestive of brain disorders, brain tumors, or metabolic or neurodegenerative diseases of rapid progression.
* Presence of acute and clinically significant diseases as assessed by a medical investigator, such as kidney, liver, urinary, bowel, or respiratory infections.
* Presence of known chronic and clinically significant diseases as assessed by a medical investigator and which may interfere with participation in the trial or pose safety risks for the participant.
* History of liver, kidney, lung, hematological, heart, or psychiatric diseases that may affect the volunteers' health or participation in the trial.
* Hypotension or hypertension with any etiology and requiring pharmacological management.
* History of surgeries that may affect the volunteers' health and/or participation in the trial.
* Regular or intermittent use of marijuana over the 60 days preceding the baseline assessment.
* Regular or intermittent treatment with CBD over the 60 days preceding the baseline assessment.
* History of allergies or idiosyncratic reactions to Cannabis sativa derivatives or components of the pharmaceutical formulation.
* Clinically significant ECG alterations as judged by a medical investigator.
* Participation in other clinical trials within less than 3 months before the baseline assessment.
* Donation or loss of 450 mL or more of blood within 90 days before the baseline assessment.
* Impaired liver function: AST, ALP, alkaline phosphatase and γGT values more than 3 times above the upper limit of the reference value. Results of γGT values 3 times above the upper limit will only be accepted if attributable to liver enzymatic induction caused by concomitant treatment with AEDs and with levels of other liver enzymes lower than 3 times the upper limit of the reference range.
* Participants with clinically significant discrepancies from the reference ranges of the following laboratory tests: creatinine clearance < 50 ml/min, platelets < 100.000/μL, and neutrophils < 1.800/μL.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2024-07-10 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Frequency of epileptic seizures | 17 th week

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade de Pesquisa Clínica HCRP-USP, Ribeirão Preto, São Paulo, Brazil